## Title: Mobile Tablet Education to Advance Caregiver Health

NCT #: NCT03417219

March 3, 2014

- **2.A.3.g. Study Measures.** *Zarit Burden Interview (ZBI)* [1]. Several versions of the ZBI have been used successfully as outcome measures in interventions for dementia caregivers [2, 3]. *Center for Epidemiological Studies-Depression (CES-D)* [4]. The CES-D is frequently used to assess depression in dementia caregivers and has been shown to be sensitive to changes in caregiver depression post intervention [5]. *Perceived Stress Scale (PSS)* [6]. The PSS has been used successfully to measure perceived stress in dementia caregivers [7]. *Global Deterioration Scale (GDS)* [8]. The GDS is a semi-structured rating of functional status in degenerative dementia. It has been successfully used in prior studies of dementia caregiver intervention with adequate reliability [9]. *Telephone Cognitive Screen (T-CogS)* [10]. The T-CogS is a brief mental status examination designed to be administered over the telephone. Scores on the T-CogS strongly correlate with MMSE scores (r = 0.88, p < 0.001) [11]. An exclusion cutoff score of < 20 on the T-CogS is chosen to match a MMSE cutoff of < 23 [12]. *Caregiver Interview*. All caregivers will also be administered a structured interview to ascertain information on levels of socialization and pleasurable activity participation.
- **2.A.3.h. Data Management.** Integrity of data collection, scoring, and entry/verification will be overseen by the MIRECC Data Analyst/Database Manager and the PI.
- **2.A.3.i.** Statistical Analyses. While the proposed project is designed to assess study feasibility, to test the hypotheses outlined in the Specific Aims (Section 2) we will use mixed-effects modeling to fully utilize outcome data measured over time (baseline and follow-up assessments) and to better handle missing outcome information in line with the intention to treat principle. Dr. Jo will serve as a statistical consultant, given her expertise in clinical trial and mixed modeling methodologies.
- 1. Zarit, S., *The hidden victims of Alzheimer's disease: Families under stress.* 1985: NYU Press.
- 2. Belle, S.H., L. Burgio, R. Burns, D. Coon, S.J. Czaja, D. Gallagher-Thompson, L.N. Gitlin, J. Klinger, K.M. Koepke, C.C. Lee, J. Martindale-Adams, L. Nichols, R. Schulz, S. Stahl, A. Stevens, L. Winter, and S. Zhang, *Enhancing the quality of life of dementia caregivers from different ethnic or racial groups: a randomized, controlled trial.* Ann Intern Med, 2006. **145**(10): p. 727-38.
- 3. Nichols, L.O., J. Martindale-Adams, R. Burns, M.J. Graney, and J. Zuber, *Translation of a dementia caregiver support program in a health care system--REACH VA.* Arch Intern Med, 2011. **171**(4): p. 353-9.
- 4. Radloff, L.S., *The CES-D Scale: A Self-Report Depression Scale for Research in the General Population.* Applied Psychological Measurement, 1977. **1**(3): p. 385-401.
- 5. Pinquart, M. and S. Sörensen, *Differences between caregivers and noncaregivers in psychological health and physical health: a meta-analysis.* Psychology and aging, 2003. **18**(2): p. 250.
- 6. Cohen, S., T. Kamarck, and R. Mermelstein, *A global measure of perceived stress*. J Health Soc Behav, 1983. **24**(4): p. 385-96.
- 7. Gallagher-Thompson, D., J.O. Brooks, 3rd, D. Bliwise, J. Leader, and J.A. Yesavage, *The relations among caregiver stress, "sundowning" symptoms, and cognitive decline in Alzheimer's disease.* J Am Geriatr Soc, 1992. **40**(8): p. 807-10.
- 8. Reisberg, B., S.H. Ferris, M.J. de Leon, and T. Crook, *The Global Deterioration Scale for assessment of primary degenerative dementia*. Am J Psychiatry, 1982. **139**(9): p. 1136-9

- 9. Mittelman, M.S., W.E. Haley, O.J. Clay, and D.L. Roth, *Improving caregiver well-being delays nursing home placement of patients with Alzheimer disease.* Neurology, 2006. **67**(9): p. 1592-9.
- 10. Roccaforte, W.H., W.J. Burke, B.L. Bayer, and S.P. Wengel, *Validation of a telephone version of the mini-mental state examination*. J Am Geriatr Soc, 1992. **40**(7): p. 697-702.
- 11. Newkirk, L.A., J.M. Kim, J.M. Thompson, J.R. Tinklenberg, J.A. Yesavage, and J.L. Taylor, *Validation of a 26-point telephone version of the Mini-Mental State Examination.* J Geriatr Psychiatry Neurol, 2004. **17**(2): p. 81-7.
- 12. Folstein, M.F., S.E. Folstein, and P.R. McHugh, "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res, 1975. **12**(3): p. 189-98.